CLINICAL TRIAL: NCT05857059
Title: Misoprostol for Induction of Labor in Obese Women: Comparison Between 25 and 50 mcg Oral Administration - a Randomized Trial
Brief Title: Misoprostol for Induction of Labor in Obese Women: Comparison Between 25 and 50 mcg Oral Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Iolanda Ferreira, Assistente Hospitalar, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUC-151-17
Record Dates: First submitted 2023-04-06; First posted 2023-05-12 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Labor, Induced; Obesity; Pregnancy; Cesarean Section
MeSH Terms: conditions — Obesity | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Pregnant women seen at the obstetric clinic of Maternidade Daniel de Matos, with a first trimester ultrasound pregnancy dating at our institution; with a maternal BMI measurement in the first trimester ≥ 30 kg/m2 and with a maternal or obstetric indication for IOL, who agreed to participate in the study. They will be randomized into two groups: one will consist of pregnant women undergoing the basic IOL protocol of Maternidade Daniel de Matos (oral misoprostol 25µcg every 2 hours); the other will be submitted to a 50µcg dosage every 2 hours, maximum of 7 doses per day (maximum 2 days). The pregnant woman will have a choice of an envelope, which will be her group assignment and will be coded until the end of the trial.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol 25 mcg (Active Comparator): Participants received misoprostol 25 mcg every 2 hours until the active stage of labour was attained or failed induction was diagnosed
  Interventions: Drug: Misoprostol 25 mcg
- Misoprostol 50 mcg (Experimental): Participants received misoprostol 25 mcg matching misoprostol 50 mcg every 2 hours until the active stage of labour was attained or failed induction was diagnosed
  Interventions: Drug: Misoprostol 50 mcg

INTERVENTIONS:
Drug: Misoprostol 25 mcg — Misoprostol 50 mcg every 2 hours
  Arms: Misoprostol 25 mcg
Drug: Misoprostol 50 mcg — Misoprostol 50 mcg every 2 hours
  Arms: Misoprostol 50 mcg

SUMMARY:
In recent decades, obesity has become a prevalent issue in Portugal, with 38.6% and 13.8% of the population being overweight or obese, respectively. Obese pregnant women have a higher rate of obstetric complications, including hypertensive complications, gestational diabetes and fetal macrosomia, leading to increased induction of labor (IOL) and cesarean section (CS) rates. To determine the effect of increasing oral misoprostol dose on CS rate in obese pregnant women undergoing IOL, a randomized controlled trial with a sample size of 114 cases in each group was calculated to detect a 15% difference in CS rate. The primary objective is to determine the effect of increasing oral misoprostol dose, with secondary goals being to compare successful IOL rates and their relationship with oral misoprostol dose, as well as to evaluate tolerability and side effects in relation to different doses of oral misoprostol.

DETAILED DESCRIPTION:
The prevalence of obesity has increased dramatically in recent decades, with implications for women of reproductive age and changes in obstetric and perinatal outcomes. In Portugal, it is estimated that 38.6 per cent and 13.8 per cent of the population are overweight or obese, respectively. Compared with women of normal weight, obese pregnant women have a higher rate of obstetric complications. These include hypertensive complications, gestational diabetes and fetal macrosomia. These factors lead to an increased need for IOL before the end of the pregnancy and, consequently, to a reduced degree of cervical dilatation prior to IOL. In addition, the above-mentioned co-morbidities are associated with a higher rate of CS. For all these reasons, obese women have higher IOL and CS rates. The literature also confirms that the degree of obesity is directly related to IOL failure. In some studies, the rate of failed induction is 20.2% and 24.2% in women with obesity grades I and II, respectively. However, few studies have been conducted to determine which IOL agents most commonly induce vaginal labour in obese women, and no studies have defined the most appropriate dose for maternal BMI.

This study provides a breakthrough in understanding the mechanism of labour and response to misoprostol in obese women, as there is a lack of prospective human studies in this area.

Sample size calculation was based on CS rate in obese versus non-obese groups as the primary outcome. According to previous studies, a 22% CS rate in non-obese pregnant women undergoing IOL was calculated, with a between-groups difference of 15% on CS rates being considered clinically significant. Therefore, we set the power at 80%, the alpha error at 0.05 and the ratio of the two study groups at 1:1. Accordingly, 114 cases were needed in each group to detect 15% difference in CS rate.

Primary objective: To determine the effect of increasing oral misoprostol dose on CS rate in obese pregnant women undergoing IOL.

Secondary goals: Comparison of successful IOL rates and their relationship with oral misoprostol dose. Evaluation of tolerability and side effects in relation to different doses of oral misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/m2 recorded based on maternal weight at preconception or in the first trimester
* Singleton live gestation with vertex presentation
* Pregnancies followed in our institution with sonographic confirmation of gestational age in the first trimester
* Obstetrical indication for labor induction
* Bishop score of <5 at the time of induction of labor

Exclusion Criteria:

* Underweight and normal weight women (BMI <30 kg/m2)
* Known hypersensitivity to prostaglandins
* Preterm gestations (< 37 weeks)
* Multiple gestation
* Women who cannot give their informed consent
* Contraindications for vaginal delivery
* Previous c-section or uterine scar due to previous gynecological surgery
* Maternal or fetal pathology (for example: fetal indications: non-reassuring fetal status - intra-uterine growth restriction with abnormal umbilical doppler, abnormal fetal cardiac rhythm; stillbirth; or maternal/pregnancy related indications such as placenta previa)

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 228 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Cesarean section rates | Up to 3 days after first misoprostol intake until delivery (vaginal or cesarean section)
  Calculation in percentage. An average of 22% cesarean section rate in non-obese pregnant women undergoing IOL was determined, with a between-groups difference of 15% on cesarean section rates being considered clinically significant.
Indication for cesarean section | Delivery
  The American College of Obstetricians and Gynecologists (ACOG) and the Society for Maternal-Fetal Medicine guidelines for caesarean section indications are used. When a caesarean section is performed, it will be classified in mutually exclusive categories. These are:
  First stage labor dystocia: Yes/No Second stage labor dystocia: Yes/No Abnormal or indeterminate fetal heart rate tracing: Yes/No Failed induction: Yes/No

SECONDARY OUTCOMES:
Rate of vaginal delivery within 24 hours | Time of first misoprostol intake until vaginal delivery
  Percentage of eutocic or instrumental deliveries that occured within a 24h of the first misoprostol intake
Time interval from the first dose of misoprostol to vaginal delivery | Time of first misoprostol intake until vaginal delivery
  Median time in hours
Rate of instrumental delivery | Delivery
  Percentage of vaginal deliveries that need instrumentation with ventouse or forceps
Time interval from the first dose of misoprostol to cesarean section delivery | Time of first misoprostol intake until cesarean section delivery
  Median time in hours
Incidence of misoprostol adverse effects | Time of first misoprostol intake until vaginal or cesarean section delivery
  Tachysystole (defined as at least six uterine contractions in 10 minutes for two consecutive 10-minute periods) and hyperstimulation (defined as the presence of tachysystole or a prolonged uterine contraction lasting 2 or more minutes associated with fetal heart rate abnormalities) will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Iolanda João Mora Cruz de Freitas Ferreira, Coimbra, Portugal